CLINICAL TRIAL: NCT03207399
Title: Lung Transplantation in Chronic HCV Infection With Post Transplant EPCLUSA Treatment: A Pilot Feasibility and Efficacy Study
Brief Title: Lung Transplantation in Chronic HCV Infection With Post Transplant EPCLUSA Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment terminated due to not having any other eligible participants.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00074361
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C, Chronic; Lung Transplant
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epclusa (Other): Epclusa (sofosbuvir 400mg/velpatasvir 100mg) 1 tablet oral or via tube daily for 12 weeks, taken with or without food.
  Interventions: Drug: Epclusa

INTERVENTIONS:
Drug: Epclusa — Patients will be treated with this drug for 12 weeks post lung transplant.

SUMMARY:
The purpose of this study is to evaluate whether treatment with Epclusa (sofosbuvir/velpatasvir) after lung transplantation in individuals with chronic hepatitis C infection is feasible, safe and effective at curing HCV.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA >= 10^3 IU/ml at screening
* Chronic HCV infection, defined as positive HCV antibody and/or HCV RNA more than 6 months prior to screening
* HCV Genotype 1, 2, 3, 4, 5 or 6
* Otherwise eligible for lung transplant at study site

Exclusion Criteria:

* Age <18
* Treatment with any of the following agents:

  * Amiodarone. Subjects previously treated with amiodarone must have stopped the amiodarone at least 60 days prior to day 1 SOF/VEL
  * Carbamazepine, phenytoin, phenobarbital, oxcarbazepine
  * Rifabutin, rifampin or rifapentine
  * HIV regimens containing tenofovir or tipranavir/ritonavir
  * St John's wort
  * PPIs, including: Omeprazole, pantoprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole
  * Modafinil
* Have any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with subject treatment, assessment or compliance
* Hepatitis B surface antigen positive
* History of hepatic encephalopathy or variceal hemorrhage
* Abnormal hematological and biochemical parameters, including:

  * Hemoglobin <8g/dL
  * Platelets <= 50,000/mm^3
  * ALT (alanine aminotransferase), AST (aspartase aminotransferase) or alkaline phosphatase >=10 times ULN
  * Total bilirubin >3mg/dL
  * Severe renal impairment, ie creatinine clearance (CrCl) <30mL/min
* Pregnant women or women planning to become pregnant
* Women or are breastfeeding
* Active or recent history (<=1 year) of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Mohamedaly, MD, Principal Investigator — Duke Heath
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epclusa
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response 12 Weeks (SVR 12) in Those Treated With EPCLUSA.
Description: Sustained Virologic Response 12 weeks (SVR 12) in those treated with EPCLUSA.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Number of Patients That Reported an Adverse Event Resulting in Discontinuation of EPCLUSA
Description: Adverse events resulting in discontinuation of EPCLUSA
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Number of Patients Eligible for EPCLUSA Treatment
Description: Eligibility for EPCLUSA treatment within 12 months of lung transplant
Time Frame: within 12 months of lung transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Change in Serum HCV RNA Levels
Description: Serum HCV RNA levels at 12-, 24-, and 48-weeks after initiation of EPCLUSA
Time Frame: 12, 24, and 48 weeks after initiation of EPCLUSA
Measure: Number; unit: IU/mL
Arm/Group | Epclusa
Number analyzed (Participants) | 1
IU/mL
  Week 12 | NA — HCV RNA value fell below the level of detection.
  Week 24 | NA — HCV RNA value fell below the level of detection.
  Week 48 | NA — HCV RNA value fell below the level of detection.

5. Secondary Outcome: Number of Participants With Adverse Events Requiring Temporary Interruption of EPCLUSA Therapy
Description: Adverse events requiring temporary interruption in EPCLUSA therapy
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Patient Survival
Description: 90-day post transplant patient survival
Time Frame: 90 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 1

7. Secondary Outcome: Patient Survival
Description: 1 year post transplant patient survival
Time Frame: 1 year post-tranplant
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 1

8. Secondary Outcome: Patient Survival
Description: 90-day post transplant patient survival in recipients of HCV NAT positive donor organ
Time Frame: 90 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 1

9. Secondary Outcome: Patient Survival
Description: 1 year post transplant patient survival in recipients of HCV NAT positive donor organ
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Epclusa
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Epclusa
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03207399/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03207399/ICF_001.pdf